CLINICAL TRIAL: NCT05094440
Title: Feasibility, Acceptability, and Efficacy of a Dialectical Behavioral Therapy Digital Health Solution in the CAMH Rainbow/COMPASS Service
Brief Title: A Dialectical Behavioral Therapy Digital Health Solution for Outpatients Seeking Support for Substance Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University of Missouri, St. Louis (Other)
Responsible Party: Principal Investigator, Lena Quilty, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 016/2021
Record Dates: First submitted 2021-10-14; First posted 2021-10-26 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Alcohol Use Disorder; Substance Use Disorders
Keywords: dialectical behavior therapy, digital health
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment (Experimental): Pocket Skills is a dialectical behavior therapy skills training (DBT-ST) webapp that includes video lessons, an interactive chatbot AI coach, and in-app exercises to practice DBT skills. The delivery of the app intervention will be primarily monitored for one month, but followed for up to 3 months, and will be supplemented with a walk through manual and links to DBT worksheets. The intervention will be delivered in conjunction with treatment as usual which includes standard psychosocial care (e.g., assessments, group, and individual programming) as part of the Addictions Program or greater community.
  Interventions: Behavioral: Dialectical behavioral therapy skills training (DBT-ST)
- Waitlist and Delayed Treatment (Active Comparator): Waitlist control whereby outpatients or members of the community will wait 1 month (4 weeks) to receive the intervention and then receive the Pocket Skills webapp for the subsequent 2 months (8 weeks). The waitlist period and subsequent intervention will be delivered in conjunction with treatment as usual which includes standard psychosocial care (e.g., assessments, group, and individual programming) as part of the Addictions Program.
  Interventions: Behavioral: Dialectical behavioral therapy skills training (DBT-ST)

INTERVENTIONS:
Behavioral: Dialectical behavioral therapy skills training (DBT-ST) — Pocket Skills is a dialectical behavior therapy skills training (DBT-ST) webapp that includes video lessons, an interactive chatbot AI coach, and in-app exercises to practice DBT skills. The delivery of the app will occur primarily over 1 month, followed by 2 months of follow-up, and will be supplemented with a walk through manual and links to DBT worksheets.
  Other Names: Pocket Skills

SUMMARY:
The purpose of this study is to compare the feasibility, acceptability, and efficacy of a dialectical behavior therapy skills training webapp known as "Pocket Skills" in outpatients and community members seeking treatment for substance use, across those who receive immediate versus delayed access to the intervention (e.g., a waitlist control condition).

DETAILED DESCRIPTION:
Seventy adult outpatients and community members seeking treatment for substance use from the Centre for Addiction and Mental Health Addictions Program will be randomized to receive immediate or delayed (1 month) access to a web-based DBT skills training intervention called Pocket Skills in addition to standard care. Participants will complete interviews and questionnaires at baseline. Following baseline, participants complete questionnaires at months 1, 2, and 3 months. Measures will assess alcohol and drug consumption, substance use disorder symptoms, and other clinical features.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age
2. Fluency in English
3. Understanding and willingness to comply with study requirements
4. Referred to Addictions Program at CAMH or seeking treatment from the community and currently waiting for psychosocial services
5. Smartphone, tablet, or computer with access to the Internet
6. Reports at least "contemplation" levels of wanting to reduce substance use
7. Use of target substance in past month
8. Alcohol or substance use disorder in the past year

Exclusion Criteria:

1. Any known practical factor that would preclude participation (e.g., extended absences)
2. Untreated or unstable severe psychiatric or medical disorder that precludes participation in the study (e.g., acute suicidality, untreated psychosis)
3. Participation in another treatment/intervention study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Severity of Dependence Scale | 30 days
  Level of dependence on most problematic substance over past 30 days. Minimum score: 0, maximum score 15. Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (Depression Subscale; PHQ-9) | 14 days
  Level of depressive symptoms over the past 14 days. Minimum score: 0, maximum score 27. Higher scores mean worse outcome.
Generalized Anxiety Disorder-7 (GAD-7) Scale | 14 days
  Level of generalized anxiety symptoms over the past 14 days. Minimum score: 0, maximum score 21. Higher scores mean worse outcome.
Difficulties in Emotion Regulation Scale, Short Form (DERS-SF; Kaufmann et al., 2015) | 30 days
  Level of emotion dysregulation or the difficulty in changing unwanted emotions effectively in the past month. Minimum score: 18, maximum score 90. Higher scores mean worse outcome.
WHO Disability Assessment Schedule Short Form (WHODAS 2.0) | 30 days
  Level of functional disability in the past month. Minimum score: 0, maximum score 48. Higher scores mean worse outcome.
Mindful Attention and Awareness Scale (MAAS) | 30 days
  Measure of core mindfulness skills around awareness and acceptance, over the past month. Minimum score: 0, maximum score 6 (mean score on 15 items). Higher scores indicate more positive outcome (e.g., more mindful awareness).
Suicidal Behaviors Questionnaire, Revised (SBQ-R; Osman et al., 2001) | 30 days
  Measure of suicidal ideation and behaviors over the past month. Minimum score: 3, maximum score: 18. Higher scores indicate worse outcome.
Risky, Impulsive, and Self-Destructive Questionnaire (RISQ) | 30 days
  Measure of risky and impulsive behavior, past month. Only subscales pertaining to sexual behavior and general reckless behavior will be used. Minimum score: 0, Maximum score: 40. Higher scores indicate worse outcome (e.g., more impulsive and/or risky behaviors)
NIDA Assist | 30 days
  Assesses the frequency of non-alcohol substance use over the past month. Minimum score per item: never used substance; maximum score per item: used substance daily or almost daily. Higher scores indicate worse outcome (e.g., more substance use).
Daily Drinking Questionnaire (DDQ) | 30 days
  Assesses the frequency and quantity of alcohol use and binge drinking episodes over the past month. Minimum score: no alcoholic drinks on specific day; Maximum score: 15+ drinks on a specific day. Higher scores indicate worse outcome (E.g., more alcoholic drinks consumed).

OTHER OUTCOMES:
Treatment Acceptability Questionnaire (TAQ; Hunsley, 1992) | 8 weeks
  Whether or not the treatment is seen as acceptable and helpful with respect to current symptoms/problems. Minimum score: 6, maximum score: 42. Higher scores indicate better treatment acceptability and positive perceptions of the treatment.
Credibility/Expectancy Questionnaire (CEQ; Devilly & Borkovec, 2000) | 30 days
  Measure of treatment credibility and expectancy for interventions. Minimum score: 4; Maximum score: 56; Higher scores mean participants perceive the intervention to provide expected benefits and/or improvements.

CONTACTS AND LOCATIONS:
Overall Officials: Lena C. Quilty, Ph.D., Principal Investigator — Campbell Family Mental Health Research Institute, CAMH
Locations (1):
- Campbell Family Mental Health Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daros AR, Guimond TH, Yager C, Palermo EH, Wilks CR, Quilty LC. Feasibility, Acceptability, and Potential Efficacy of a Self-Guided Internet-Delivered Dialectical Behavior Therapy Intervention for Substance Use Disorders: Randomized Controlled Trial. JMIR Ment Health. 2024 Jan 16;11:e50399. doi: 10.2196/50399. PMID 38227362
- See also: Information about research at the Centre for Addiction and Mental Health — http://camh.ca/research